CLINICAL TRIAL: NCT03717129
Title: Bioequivalence of Crushed and Whole Genvoya Tablets (Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Fumarate)
Brief Title: Analysis of Crushed and Whole Tablet Genvoya
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB00110315; IN-US-292-4089 (Other Grant/Funding Number: Gilead)
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — elvitegravir; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Genvoya Oral dose (Active Comparator): Single observed oral dose of Genvoya whole tablet
  Interventions: Drug: Genvoya Oral dose
- Genvoya Crushed Dose (Experimental): Single observed oral dose of Genvoya crushed tablet
  Interventions: Drug: Genvoya Crushed Dose

INTERVENTIONS:
Drug: Genvoya Oral dose — Single Genvoya oral dose directly observed
  Other Names: elvitegravir/cobicistat/emtricitabine/ tenofovir alafenamide
  Arms: Genvoya Oral dose
Drug: Genvoya Crushed Dose — Single Genvoya crushed tablet in water directly observed
  Other Names: elvitegravir/cobicistat/emtricitabine/ tenofovir alafenamide
  Arms: Genvoya Crushed Dose

SUMMARY:
Step-wise, two sequential, single-dose, bioequivalence study in 12 healthy volunteers to determine whether crushed Genvoya tablet is bioequivalent to whole Genvoya tablet. The first study sequence will involve a directly observed single dose of the fixed dose formulation of whole Genvoya tablet, with semi-intensive pharmacokinetic serum sampling at time points following the dose. After a washout period of seven days, subjects will then receive a directly observed single dose of a crushed tablet of Genvoya with subsequent semi-intensive pharmacokinetic serum sampling.

DETAILED DESCRIPTION:
Genvoya, a fixed-dose combination of the two Nucleoside Reverse Transcriptase Inhibitors (NRTI) emtricitabine (FTC) 200mg and tenofovir alafenamide (TAF) 10mg, with the integrase inhibitor elvitegravir (EVG) and the boosting agent cobicistat (COBI), is FDA approved for the treatment of HIV-infected patients.

Despite the availability of Genvoya allowing for a single tablet fixed-dose combination and once-daily dosing, a substantial number of individuals living with HIV suffer from pill aversion, dysphagia, odynophagia, or problems swallowing oral regimens, all of which can contribute to non-adherence. These observations are especially important because non-adherence to antiretroviral (ARV) medications is highly prevalent and associated with decreased survival. Non-adherence has been estimated at 55% in North American pooled cohorts, and is a vital public health concern, as it leads to treatment failure and transmission of drug-resistant virus.

Many clinical scenarios make the administration of crushed tablets desirable as a potential strategy to overcome pill aversion. However, there is a theoretical concern that the systemic absorption of the active ingredients of tablets may be altered by crushing the pills. In fact, pharmacokinetic and bioequivalence data are lacking for most antiretroviral fixed-dose combinations used in the treatment of HIV-infected patients. It is therefore of substantial practical and clinical interest to know whether antiretroviral combinations such as Genvoya can be taken in crushed form with bioequivalence to whole tablet form.

This is a step-wise bioequivalence single-dose and two sequential design study in healthy volunteers to evaluate the combination Genvoya to provide this critical information.

Primary Objective: To investigate the bioequivalence of oral single whole tablet and crushed tablet of Genvoya in healthy volunteers, by characterizing the serum Area Under the Curve 0 to infinity (AUC0-∞) and Cmax of EVG, COBI, FTC, and TAF in plasma, after single doses of whole tablet and crushed tablet of this fixed dose antiretroviral combination in healthy volunteers.

Primary Endpoint:Ratio of serum AUC0-∞ and ratio of Cmax in plasma of EVG, COBI, FTC, and TAF in healthy volunteers after two different dosage forms (whole and crushed tablets).

Secondary Endpoints(s): Ratio of Tmax in plasma of EVG, COBI, FTC, and TAF in healthy volunteers after two different dosage forms (whole and crushed tablets).

Projected Study Design: Step-wise, two sequential, single-dose, bioequivalence study in 12 healthy volunteers. The first study sequence will involve a directly observed single dose of the fixed dose formulation of whole Genvoya tablet, with semi-intensive pharmacokinetic serum sampling at time points following the dose. After a washout period of seven days, subjects will then receive a directly observed single dose of a crushed tablet of Genvoya with subsequent semi-intensive pharmacokinetic serum sampling. Additional information about the proposed pharmacokinetic sampling time points for each of the antiretroviral components of Genvoya and safety evaluations is included in the Study Procedures Section of this proposal. The duration of the washout period of seven days between the two study sequences and proposed pharmacokinetic sampling time points, was selected for convenience and based on the antiretroviral component of Genvoya with the longest half-life (EVG).

Projected Duration of Treatment: Two directly observed doses of one table of Genvoya over two weeks (one single dose of whole and one single dose crushed Genvoya tablets, as specified in the Regimen Section of this proposal).

Study Duration: It will take 6-8 months to complete accrual and follow up of 12 subjects and an additional three months to complete the data analysis.

Regimens - Study Sequence:

Period 1: Product: Genvoya - Dose: 1 tablet PO (whole) - Frequency: Single dose Period 2: Product: Genvoya - Dose: 1 tablet PO (crushed) - Frequency: Single dose

Other Evaluations: Safety will be monitored and evaluated at pre-defined time points (screening and 2 weeks) throughout the study, and assessments will include: monitoring for adverse treatment-related events, clinical examinations with vital signs, and collection of blood for routine safety laboratory tests in accordance with the protocol [e.g. Complete Blood Count (CBC), chemistry, HIV and hepatitis B (HBV screening, pregnancy test]. Subjects will receive a single dose of Genvoya whole and crushed tablets. Pharmacokinetic assessment will be performed, with blood drawn for testing at time zero, and at selected time points after dosing with for EVG, COBI, FTC, and TAF, with more intensive sampling surrounding the evidence-based Cmax of each drug, and adequate sampling in the tail to estimate AUC with precision. Plasma will be tested for EVG, COBI, FTC and TAF concentrations using a validated high-performance liquid chromatography- mass spectroscopy (HPLC-MS) assay. The ARV components of Genvoya will be sampled as follows:

EVG -10 time points: 0, 1, 2, 3, 4, 9, 12, 24, 48, 72 hours COBI -11 time points: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 18, 24 hours FTC-14 time points: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48, 72 hours TAF-10 time points: (0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6 hours

To determine serum pharmacokinetic parameters of EVG, COBI, FTC, and TAF the Phoenix WinNonLin non-linear curve-fitting software (V 6.4; Pharsight, Mountain View, CA) will be employed using standard non-compartmental analytic methods. Pharmacokinetic parameters calculated will include area under the plasma concentration-time curve from 0 to τ (AUCτ, calculated using the linear trapezoidal rule); the maximum EVG, COBI, FTC, and TAF concentrations in serum after one dose (Cmax); and the time to maximum observed drug concentrations in serum (Tmax).

Hypothesis: there will be a 90% confidence interval between 0.8 and 1.25 for the ratio of Area Under the Curve for the whole tablet (AUCwhole): Area Under the Curve for the crushed tablet (AUCcrushed); and the ratio of Maximum Concentration whole tablet (Cmaxwhole): Maximum Concentration crushed tablet (Cmaxcrushed), for the four antiretroviral components of Genvoya: EVG, COBI, FTC, and TAF.

An equivalence approach with no-effect boundaries of 80 to 125% will be employed, in accordance with the FDA guidance on bioequivalence studies, which define bioequivalence as "the absence of a significant difference in the rate and extent to which the active moiety becomes available at the site of action when administered at the same molar dose under similar conditions.

In order to test the primary hypothesis, log-transformed AUCτ and Cmax after a single dose for crushed versus whole tablets will be compared. The adjusted mean differences and ratios will be estimated and the 90% confidence intervals calculated. In the case of AUCτ and Cmax, the estimated differences and confidence limits will be exponentiated in order to compare ratios between tablet forms. For Tmax, arithmetic means will be calculated, whereas for AUCτ and Cmax, geometric means will be calculated.

Statistical methods. The sample size was calculated according to the formulas for a multiplicative model. Table 2 includes sample size calculations for this proposed study. If the mean Cmax ratio or AUC ratio is 1, a sample size of 5 subjects produces a two-sided 90% confidence interval (0.952, 1.048) (i.e., a distance from the mean to the limits that is equal to 0.048, when the estimated standard deviation is 0.050). A sample size of 10 subjects produces a two-sided 90% confidence interval (0.855, 1.145) if the mean Cmax ratio or AUC ratio is 1, and the estimated standard deviation is 0.25. Assuming a dropout rate of 10%, a sample size of 12 subjects will be required required to provide 90% power to demonstrate the bioequivalence of Cmax with 90% confidence intervals (CI) of 80% and 125%

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female research participants, ≥18 years of age.
* Negative HIV-1/2 Ag/Ab serology documented within 30 days prior to study entry.
* Negative Hepatitis B surface antigen within 30 days prior to study entry.
* Ability and willingness of subject to provide a signed informed consent and comply with study requirements.
* Negative qualitative urine pregnancy test.
* All subjects must not participate purposely in a conception process (e.g., active attempt to impregnate, sperm donation, or in vitro fertilization). If participating in sexual activity that could lead to pregnancy subjects must take every precaution to avoid risk of pregnancy by using a reliable contraception for the duration of the study therapy (e.g., condoms, hormonal, barrier).
* Laboratory values and physical examination as judged by the principal investigator to be safe to participate including normal renal function.
* Good peripheral venous access for proposed pharmacokinetic sampling.
* Willingness and ability to take oral medications.

Exclusion Criteria:

* History of chronic or acute medical conditions that in the opinion of the investigator would jeopardize safety of subjects participating in this study.
* Known or suspected hypersensitivity to the components of Genvoya.
* Use of prescription or over-the-counter medications, including agents containing polyvalent cations (e.g., Mg, Al, Fe, or Ca), or any other drugs that in the opinion of the investigator could interfere with the pharmacokinetics of any of the ARV components of Genvoya within 2 weeks prior to either study dose.
* Pregnant or breast feeding.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Hospitalization or therapy for serious illness within 30 days prior to study entry as judged by the investigator.
* Participation in any investigational drug study within 30 days prior to study entry that in the opinion of the investigator would preclude study participation.
* Taking any medication listed in the package insert that is contraindicated with Genvoya.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Principal Investigator — JHU
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andrade A, Fuchs EJ, Marzinke MA, Abdul Massih S, Breakey J, Beselman S, McNicholl I, Hendrix CW. EVG/COBI/FTC/TAF Bioequivalence Comparing Whole Tablets with Tablets Dissolved in Tap Water. AIDS Res Hum Retroviruses. 2023 Jan;39(1):38-43. doi: 10.1089/AID.2022.0085. Epub 2022 Dec 22. PMID 36301928

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a cross-over study where participants acted as their own controls. All participants received Genvoya oral first, and then crossed over to Genvoya crushed after a 2-week washout period.
Period: Genvoya Oral Dose (1 Week)
Arm/Group | Genvoya Oral Dose
Started | 12
Completed | 12
Not Completed | 0
Period: Washout (2 Weeks)
Arm/Group | Genvoya Oral Dose
Started | 12
Completed | 12
Not Completed | 0
Period: Genvoya Crushed Dose (1 Week)
Arm/Group | Genvoya Oral Dose
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants received Genvoya Oral Dose and then, after a washout period, received Genvoya Crushed Dose.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From 0 to Infinity (AUC0-∞) for EVG
Description: AUC 0 to Infinity for Elvitegravir (ng*h/mL)
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
Number analyzed (Participants) | 12 | 12
ng*h/mL | 24219 (6074) | 26948 (5955)

2. Primary Outcome: AUC0-∞ for COBI
Description: AUC 0 to Infinity for Cobicistat (ng*h/mL)
Time Frame: 72 hours
Population: Data was not collected for this outcome
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: AUC0-∞ for FTC
Description: AUC 0 to Infinity for Emtricitabine (ng*h/mL)
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
Number analyzed (Participants) | 12 | 12
ng*h/mL | 11603 (2296) | 10969 (1818)

4. Primary Outcome: AUC0-∞ for Tenofovir (TFV)
Description: AUC 0 to Infinity for TFV (ng*h/mL)
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
Number analyzed (Participants) | 12 | 12
ng*h/mL | 253 (47) | 241 (46)

5. Secondary Outcome: EVG Cmax
Description: Maximum Plasma Concentration (Cmax) for Elvitegravir (ng/mL)
Time Frame: 72 Hr
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
Number analyzed (Participants) | 12 | 12
ng/mL | 1650 (371) | 1946 (545)

6. Secondary Outcome: FTC Cmax
Description: Maximum Plasma Concentration (Cmax) for Emtricitabine (ng/mL)
Time Frame: 72 hr
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
Number analyzed (Participants) | 12 | 12
ng/mL | 2095 (445) | 1968 (481)

7. Secondary Outcome: TFV Cmax
Description: Maximum Plasma Concentration (Cmax) for Tenofovir (ng/mL)
Time Frame: 72 hr
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
Number analyzed (Participants) | 12 | 12
ng/mL | 11 (4.1) | 9.5 (2.3)

8. Secondary Outcome: EVG Half-life
Description: Terminal elimination half-life for EVG (hours).
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
Number analyzed (Participants) | 12 | 12
hours | 5 (0.52) | 5.1 (0.56)

9. Secondary Outcome: COBI Half-life
Description: Terminal elimination half-life for COBI (hours)
Time Frame: 72 hours
Population: Data was not collected for this outcome.
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: FTC Half-life
Description: Terminal elimination half-life for FTC (hours).
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
Number analyzed (Participants) | 12 | 12
hours | 15.2 (5.2) | 16.1 (3.9)

11. Secondary Outcome: TFV Half-life
Description: Terminal elimination half-life for TFV (hours).
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
Number analyzed (Participants) | 12 | 12
hours | 42.5 (6.7) | 40.7 (13.9)

ADVERSE EVENTS:
Time Frame: Adverse event were collected for the duration of the study up until the last safety visit, which is 7 days + 3 days following the direct observed dose of Genvoya for a safety study visit, up to one month on average.
Arm/Group | Genvoya Oral Dose | Genvoya Crushed Dose
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT03717129/Prot_SAP_002.pdf
  • Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT03717129/ICF_003.pdf